CLINICAL TRIAL: NCT00003931
Title: Assessment of the Partial Tandem Duplication of ALL1 (MLL) in Patients With Acute Myeloid Leukemia- A CALGB Leukemia Tissue Bank Project
Brief Title: Diagnostic Study of Gene Alterations in Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9769; U10CA031946 (NIH); CLB-9769; CDR0000067123 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-08-20 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood or bone marrow samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- blood or bone marrow samples: All samples are obtained from specimens collected on CALGB-9665. No additional blood or bone marrow samples are collected CALGB-9769.
  Samples are examined by Southern blot analysis for gene rearrangement at 11q23. Samples showing evidence of ALL1 gene rearrangement are further analyzed by reverse transcription PCR amplification and/or cytogenetic analysis to detect partial tandem duplication of ALL1.
  Interventions: Genetic: reverse transcriptase-polymerase chain reaction

INTERVENTIONS:
Genetic: reverse transcriptase-polymerase chain reaction

SUMMARY:
RATIONALE: Diagnostic procedures, such as genetic testing, may improve the ability to detect acute myeloid leukemia and determine the extent of disease.

PURPOSE: Diagnostic study to try to detect changes in the genes of patients who have acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of partial tandem duplication of ALL1 (MLL) in patients with acute myeloid leukemia (AML).
* Determine the predictive value of partial tandem duplication of ALL1 to identify a subset of AML patients who have a short duration of complete remission.

OUTLINE: All samples are obtained from specimens collected on CALGB-9665. No additional blood or bone marrow samples are collected.

Samples are examined by Southern blot analysis for gene rearrangement at 11q23. Samples showing evidence of ALL1 gene rearrangement are further analyzed by reverse transcription PCR amplification and/or cytogenetic analysis to detect partial tandem duplication of ALL1.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior registration on protocol CALGB-9665
* Diagnosed with acute myeloid leukemia (AML)
* Treated on a CALGB AML treatment protocol
* Diagnostic bone marrow or blood specimen available

PATIENT CHARACTERISTICS:

Age:

* 15 and over

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously enrolled on CALGB-9665.
Sampling Method: Non-Probability Sample
Enrollment: 9769 (Actual)
Dates: Start 1999-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
frequency of partial tandem duplication of ALL1 (MLL) | Up to 10 years

SECONDARY OUTCOMES:
predictive value of partial tandem duplication of ALL1 | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Caligiuri, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (46):
- United States (46):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia